CLINICAL TRIAL: NCT06242756
Title: A Randomized Controlled Trial of Use Versus Non-use of Bladder Catheterization in Elective Cesarean Delivery
Brief Title: Use Versus Non-use of Bladder Catheterization in Elective Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB24-0044
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; bladder catheterization; foley
MeSH Terms: interventions — Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder catheterization (Experimental): Patients placed in the catheterized group will have an indwelling catheter placed after anesthetic has been administered. It would be removed at 12 hours post Cesarean section.
  Interventions: Procedure: Bladder catheterization
- Non-use of bladder catheterization (No Intervention): Participants in the non-catheterized group would be encouraged to empty their bladders just prior to transfer to the operating room where they will undergo surgery without an indwelling catheter.

INTERVENTIONS:
Procedure: Bladder catheterization — Patients placed in the catheterized group will have an indwelling catheter placed after anesthetic has been administered. It would be removed at 12 hours post cesarean section.
  Arms: Bladder catheterization

SUMMARY:
The goal of this randomized controlled trial is to investigate the impact of routine bladder catheterization in uncomplicated cesarean sections on hospitalization time (readiness to discharge), time to ambulation, urinary retention, development of urinary tract infections, prevention of bladder injury, operating time, and patient satisfaction.

DETAILED DESCRIPTION:
This would be a randomized controlled trial conducted on the labour and delivery and post-partum unit at a large academic site (Foothills Medical Centre) in Calgary, Alberta. Study recruitment of patients awaiting delivery via CS would occur either in participating prenatal clinics in Calgary or in obstetrical triage by a trained nurse research assistant. Participants would be randomized into either a catheterized or non-catheterized group prior to their scheduled elective CS. Allocation concealment will be ensured by using either a central computer generator for randomization if funding permits, otherwise sealed, opaque, and sequenced envelopes will be used. Since there may be potential differences in patients with increasing parity, randomization will be stratified by parity and blocked to prevent imbalance in treatment groups.

ELIGIBILITY:
Inclusion criteria:

- women who are 18 years of age or older with a singleton pregnancy presenting for an elective primary or repeat CS.

Exclusion criteria:

- diagnosis of abnormal placentation including placenta previa, vasa previa, or suspected invasive disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time at readiness for discharge post-surgery | Prior to discharge, average of 2 days postpartum
  Time at readiness for discharge post-surgery will be collected via a form that will be distributed to the postpartum nursing team.
Time to ambulation | Prior to discharge, an average of 2 days postpartum
  Time to ambulation will be collected via a form that will be distributed to the postpartum nursing team.

SECONDARY OUTCOMES:
Incidence of urinary retention | Prior to discharge, an average of 2 days postpartum
  Urinary retention will be defined based on a patient's inability to spontaneously void requiring either in-and-out catheterization or placement of an indwelling catheter during the post operative course
Incidence of urinary tract infections (UTI) requiring antibiotics in the first 4 weeks postpartum | first 4 weeks postpartum
  Incidence of urinary tract infections (UTI) requiring antibiotics in the first 4 weeks postpartum
Incidence of bladder injury in surgery | During surgery
  Incidence of bladder injury in surgery will be collected via an electronic post-operative questionnaire filled out by the operating surgeon.
Operating time | During surgery
  Operating time will be collected via an electronic post-operative questionnaire filled out by the operating surgeon.
Patient satisfaction as measured by the Maternal Satisfaction for Cesarean Section questionnaire (MSCS) | Prior to discharge, an average of 2 days postpartum
  Patients will be asked to complete the Maternal Satisfaction for Cesarean Section questionnaire at discharge. The minimum and maximum values are 7 and 154 and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L. Wood, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT06242756/Prot_SAP_000.pdf